CLINICAL TRIAL: NCT01004848
Title: Collaborations for Health Improvement in East Harlem-Project HEED
Brief Title: Effectiveness Study of Community-Based, Peer-Led Education on Weight Loss and Diabetes
Acronym: HEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: North General Hospital, New York (Other); Albert Einstein College of Medicine (Other); Union Settlement Association, New York (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 05-0463
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Pre-diabetes
Keywords: Pre-diabetes; pre-diabetic state; community-based participatory research; overweight; weight loss intervention, peer-led lifestyle education
MeSH Terms: conditions — Glucose Intolerance; Overweight

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer-Led Lifestyle Education on Weight Loss (Experimental): Project HEED (Help Educate to Eliminate Diabetes), a community-based, peer-led weight loss program for overweight adults with pre-diabetes.
  The intervention group will participate in an 8-session course held over a 10-week period. Project HEED (Help Educate to Eliminate Diabetes), led by trained peer educators, aims to help participants lose weight, thereby preventing their progression to diabetes.
  Interventions: Behavioral: Peer-Led Lifestyle Education on Weight Loss
- Delayed Intervention (Placebo Comparator): The control group will be offered the chance to participate in the 8-session course 1 year after enrollment into the trial.
  Interventions: Behavioral: Peer-Led Lifestyle Education on Weight Loss

INTERVENTIONS:
Behavioral: Peer-Led Lifestyle Education on Weight Loss — Project HEED (Help Educate to Eliminate Diabetes) is a bilingual lifestyle education program written at a 4th grade reading level, and contains simple, actionable, messages, is easily taught by lay leaders, and focuses on enhancing self-efficacy to make lifestyle changes. It consists of 8 sessions (1½ hours each) held over 10-weeks. Topics include diabetes prevention, finding and affording healthy foods, label reading, fun physical activity, planning a healthy plate, making traditional foods healthy, and portion control.
  Other Names: Project HEED

SUMMARY:
The purpose of this study is to compare the effectiveness of a peer-led community-based lifestyle intervention, versus usual care, in achieving weight loss and prevention of diabetes among overweight adults with pre-diabetes in East Harlem.

DETAILED DESCRIPTION:
Weight loss can prevent diabetes and eliminate racial and ethnic disparities in incident diabetes among overweight adults with pre-diabetes. However, proven effective interventions have not been sustained or disseminated in community settings. A community-academic partnership aims to employ community-based participatory research to conduct a randomized controlled trial to test the effectiveness of a culturally tailored, peer-led diabetes prevention intervention that promotes weight loss.

People who develop diabetes go through a period when they have "pre-diabetes". In clinical settings, overweight adults with pre-diabetes who reduce their weight by 5-10% can reduce their risk of developing diabetes by 55-60%. To date, there are no studies testing the effectiveness of peer-led, community-based programs in achieving diabetes prevention through weight loss.

We will identify and enroll 400 overweight (BMI > 25) adults with pre-diabetes in East Harlem and randomized half into a community-based, peer-led lifestyle education program that teaches simple ways to lose weight.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Residents of East Harlem or members of an East Harlem Institution in zip codes 10029, 10035, OR in the section of 10037 east of Fifth Avenue
* BMI ≥ 25 AND pre-diabetes glucose values, defined as fasting fingerstick glucose of 100-125mg/dl and/or glucose 2 hours after an oral glucose load of 140-199 mg/dl
* Able to communicate verbally to participate in a group education class
* English or Spanish speaking

Exclusion Criteria:

* < 18 years
* Previous diagnosis of diabetes
* BMI <25
* Fingerstick glucoses outside pre-diabetes level ranges
* Currently pregnant
* On medications that may raise or lower blood glucose
* Cognitive or physical impairment that would preclude comprehension of a conversation and communicating as part of a group (i.e., dementia, deafness, inability to speak)
* Self-reported terminal illness with life expectancy of less than 1 year
* Plans to relocate from New York City within one year of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol R Horowitz, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Goldfinger JZ, Arniella G, Wylie-Rosett J, Horowitz CR. Project HEAL: peer education leads to weight loss in Harlem. J Health Care Poor Underserved. 2008 Feb;19(1):180-92. doi: 10.1353/hpu.2008.0016. PMID 18263994
- [Background] Cowie CC, Rust KF, Ford ES, Eberhardt MS, Byrd-Holt DD, Li C, Williams DE, Gregg EW, Bainbridge KE, Saydah SH, Geiss LS. Full accounting of diabetes and pre-diabetes in the U.S. population in 1988-1994 and 2005-2006. Diabetes Care. 2009 Feb;32(2):287-94. doi: 10.2337/dc08-1296. Epub 2008 Nov 18. PMID 19017771
- [Background] Cowie CC, Rust KF, Byrd-Holt DD, Eberhardt MS, Flegal KM, Engelgau MM, Saydah SH, Williams DE, Geiss LS, Gregg EW. Prevalence of diabetes and impaired fasting glucose in adults in the U.S. population: National Health And Nutrition Examination Survey 1999-2002. Diabetes Care. 2006 Jun;29(6):1263-8. doi: 10.2337/dc06-0062. PMID 16732006
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Hamman RF, Wing RR, Edelstein SL, Lachin JM, Bray GA, Delahanty L, Hoskin M, Kriska AM, Mayer-Davis EJ, Pi-Sunyer X, Regensteiner J, Venditti B, Wylie-Rosett J. Effect of weight loss with lifestyle intervention on risk of diabetes. Diabetes Care. 2006 Sep;29(9):2102-7. doi: 10.2337/dc06-0560. PMID 16936160
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Biuso TJ, Butterworth S, Linden A. A conceptual framework for targeting prediabetes with lifestyle, clinical, and behavioral management interventions. Dis Manag. 2007 Feb;10(1):6-15. doi: 10.1089/dis.2006.628. PMID 17309360
- [Background] Horowitz CR, Brenner BL, Lachapelle S, Amara DA, Arniella G. Effective recruitment of minority populations through community-led strategies. Am J Prev Med. 2009 Dec;37(6 Suppl 1):S195-200. doi: 10.1016/j.amepre.2009.08.006. PMID 19896019
- [Background] Fox AM, Mann DM, Ramos MA, Kleinman LC, Horowitz CR. Barriers to physical activity in East harlem, new york. J Obes. 2012;2012:719140. doi: 10.1155/2012/719140. Epub 2012 Jul 12. PMID 22848797
- [Background] Fei K, Fox A, Horowitz CR, Lee E. Family History and Perceptions of Control over Risk for Diabetes, SGIM Supplement 2012. PMC Journal - In Process.
- [Background] Breland JY, Fox AM, Horowitz CR, Leventhal H. Applying a common-sense approach to fighting obesity. J Obes. 2012;2012:710427. doi: 10.1155/2012/710427. Epub 2012 Jun 28. PMID 22811889
- [Result] Parikh P, Simon EP, Fei K, Looker H, Goytia C, Horowitz CR. Results of a pilot diabetes prevention intervention in East Harlem, New York City: Project HEED. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S232-9. doi: 10.2105/AJPH.2009.170910. Epub 2010 Feb 10. PMID 20147680

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer-Led Lifestyle Education on Weight Loss: Project HEED (Help Educate to Eliminate Diabetes), a community-based, peer-led weight loss program for overweight adults with pre-diabetes.
  The intervention group participated in an 8-session course held over a 10-week period. Project HEED (Help Educate to Eliminate Diabetes), led by trained peer educators, aims to help participants lose weight, thereby preventing their progression to diabetes.
- Delayed Intervention: The control group was be offered the chance to participate in the 8-session course 1 year after enrollment into the trial.
Period: Overall Study
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Started | 210 | 192
Completed | 155 | 147
Not Completed | 55 | 45
Not completed — Lost to Follow-up | 55 | 45

BASELINE CHARACTERISTICS:
Groups:
- Peer-Led Lifestyle Education on Weight Loss: Project HEED (Help Educate to Eliminate Diabetes), a community-based, peer-led weight loss program for overweight adults with pre-diabetes.
  The intervention group participated in an 8-session course held over a 10-week period. Project HEED (Help Educate to Eliminate Diabetes), led by trained peer educators, aimed to help participants lose weight, thereby preventing their progression to diabetes.
- Delayed Intervention: The control group offered the chance to participate in the 8-session course 1 year after enrollment into the trial.
- Total: Total of all reporting groups
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention | Total
Number analyzed (Participants) | 210 | 192 | 402
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 186 | 170 | 356
  >=65 years | 24 | 22 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 165 | 343
  Male | 32 | 27 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 153 | 141 | 294
  Not Hispanic or Latino | 55 | 48 | 103
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 41 | 93
  White | 0 | 3 | 3
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 155 | 144 | 299

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline to 6 Months
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Delayed Intervention: The control group was offered the chance to participate in the 8-session course 1 year after enrollment into the trial.
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
pounds | -2.85 (7.42) | -1.13 (7.11)

2. Secondary Outcome: Change in Fasting Fingerstick Glucose Measurement From Baseline to 6 Months
Description: Change in sugar level as measured from fingerstick, at 6 Months as compared to Baseline
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mg/dL | -1.79 (9.41) | -0.47 (9.98)

3. Secondary Outcome: Change in Post-prandial Fingerstick Glucose From Baseline to 6 Months
Description: Change in sugar level as measured from fingerstick after a meal, at 6 Months as compared to Baseline
Time Frame: Change in 6 Months from Baseline
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mg/dL | 1.41 (26.59) | 3.85 (33.14)

4. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to 6 Months
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mmHg | -1.39 (11.84) | -1.45 (12.77)

5. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to 6 Months
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mmHg | -0.47 (8.33) | -1.07 (7.96)

6. Secondary Outcome: Waist Circumference
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
inches | -0.5 (1.99) | -0.29 (2.06)

7. Secondary Outcome: LDL Cholesterol
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mg/dl | -2.93 (18.17) | -1.18 (17.87)

8. Secondary Outcome: HDL Cholesterol
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mg/dl | 0.68 (8.26) | .029 (7.17)

9. Secondary Outcome: Total Cholesterol
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mg/dl | -2.78 (21.37) | -0.66 (20.22)

10. Secondary Outcome: Triglycerides
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
mg/dl | -0.1 (52.95) | 2.92 (57.39)

11. Secondary Outcome: HbA1c
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
percent change | 0.03 (0.0485) | 1.20 (0.0553)

12. Secondary Outcome: Energy Expenditure
Description: percent energy expenditure
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: percent expenditure/day
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
percent expenditure/day | -58.08 (1.6429) | -12.54 (0.6594)

13. Secondary Outcome: Fiber Intake
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Number analyzed (Participants) | 155 | 147
grams per day | -0.19 (0.6377) | 0.013 (0.6594)

14. Secondary Outcome: Physical Activity (Self-report)
Time Frame: 6 months
Reporting Status: Not Posted

15. Secondary Outcome: Knowledge & Attitudes About Diabetes Risk
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: not applicable - adverse events not collected
Arm/Group | Peer-Led Lifestyle Education on Weight Loss | Delayed Intervention
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes